CLINICAL TRIAL: NCT01249508
Title: A University Canteen-based Labeling Program to Promote Healthy Dietary Patterns
Brief Title: Nutrition Labeling Program to Promote Healthy Dietary Patterns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Prof. Dr. Ir. Wim Verbeke, University Ghent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: EC/2008/482
Record Dates: First submitted 2010-11-25; First posted 2010-11-29 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-12

CONDITIONS: Nutrition; Diet
MeSH Terms: interventions — Food Labeling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- implemented nutrition label (Experimental): A one-group pre-/post-design is used for the evaluation of the university canteen-based nutrition labeling program. This means that all participants of the program are exposed to the nutrition label implemented in the university canteen. The subject essentially serves as its own control based on pre-test behaviour. The nutrition label implemented is a star rating label calculated and assigned to each meal offered at the university canteens and based on the content of energy, saturated fat, sodium and fibre (expressed as vegetable portion).
  Interventions: Other: nutrition label

INTERVENTIONS:
Other: nutrition label

SUMMARY:
This study aims to evaluate a nutrition labelling program in improving university canteen customers' dietary pattern and behavioural determinants (e.g. knowledge).

DETAILED DESCRIPTION:
The increase in diet related diseases worldwide is considered to be primarily caused by a changing environment encouraging high energy intakes and a sedentary lifestyle. Examples of important environmental factors are the changing nature of the food supply, the changing socio-demographic structure of the population, the lack of nutrition information and the increasing reliance on foods consumed away from home. This evolution has driven the development of measures to encourage more healthy eating patterns. Nutrition labelling is one of those measures. Since adults and students spend approximately half their waking hours at the workplace or university, the work or study environment is believed to be an appropriate setting to assess and try to change individuals' dietary behaviour. This study aims to evaluate a nutrition labelling program in improving university canteen customers' dietary pattern and behavioural determinants (e.g. knowledge).

ELIGIBILITY:
Inclusion Criteria:

* university students and staff
* frequent university canteen customers
* willing to participate

Exclusion Criteria:

* non-frequent university canteen customers

Ages: 17 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 474 (Actual)
Dates: Start 2008-10; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
pre-label behavioural determinants of nutrition | at 1 month
  Behavioural determinants of nutrition by means of quantitative questionnaire at pre-labeling implementation phase (at 1 month).
pre-label nutrition information processing characteristics | at 1 month
  Nutrition information processing by means of quantitative questionnaire at pre-labeling implementation phase (at 1 month).
post-label behavioural determinants of nutrition | at 6 months
  Behavioural determinants of nutrition by means of quantitative questionnaire at post-labeling implementation phase (at 6 months).
post-label nutrition information processing characteristics | at 6 months
  Nutrition information processing by means of quantitative questionnaire at post-labeling implementation phase (at 6 months).
pre-label food intake records | at 1 month
  Food intake by 3-day food records at pre-labeling implementation phase (at 1 month).
post-label food intake records | at 6 months
  Food intake by 3-day food records at post-labeling implementation phase (at 6 months).

SECONDARY OUTCOMES:
socio-demographic questionnaire | at 1 month
  Socio-demographical questionnaire at pre-labeling implementation phase (at 1 month).
pre-label physical activity registration | at 1 month
  Physical activity by 3-day physical activity registrations at pre-labeling implementation phase (at 1 month).
post-label physical activity registration | at 6 months
  Physical activity by 3-day physical activity registrations at post-labeling implementation phase (at 6 months).

CONTACTS AND LOCATIONS:
Overall Officials: Wim Verbeke, PhD, Prof, Principal Investigator — University Ghent
Locations (1):
- University Ghent, Ghent, Belgium

REFERENCES:
- [Derived] Hoefkens C, Pieniak Z, Van Camp J, Verbeke W. Explaining the effects of a point-of-purchase nutrition-information intervention in university canteens: a structural equation modelling analysis. Int J Behav Nutr Phys Act. 2012 Sep 11;9:111. doi: 10.1186/1479-5868-9-111. PMID 22967195
- [Derived] Hoefkens C, Lachat C, Kolsteren P, Van Camp J, Verbeke W. Posting point-of-purchase nutrition information in university canteens does not influence meal choice and nutrient intake. Am J Clin Nutr. 2011 Aug;94(2):562-70. doi: 10.3945/ajcn.111.013417. Epub 2011 Jun 15. PMID 21677060